CLINICAL TRIAL: NCT00813800
Title: Varenicline for Smoking Cessation in Bipolar Depressed Patients: An Open-Label 12-week Feasibility Trial
Brief Title: Varenicline in Bipolar Depressed Patients
Acronym: Varenicline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mark Frye (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Mark Frye, MD, Professor of Psychiatry, College of Medicine, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-003471
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Results first posted 2012-01-30 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2011-12

CONDITIONS: Smoking; Bipolar Disorder; Depression
Keywords: Smoking; Bipolar Disorder; Depression
MeSH Terms: conditions — Smoking; Bipolar Disorder; Depression | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Varenicline (Experimental): Open-label; subjects will receive a behavioral intervention in addition to Varenicline.
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — Varenicline (Chantix®, Pfizer) is an oral medication with a recommended dosage of 0.5 mg once daily for 3 days, increasing to 0.5 mg twice daily for days 4-7, and then to the maintenance dose of 1 mg twice daily for the 12 weeks of treatment.
  Other Names: Chantix

SUMMARY:
Patients with bipolar disorder have one of the highest rates of nicotine dependence and one of the lowest quit rates. Varenicline has been shown in previous trials to be effective for smoking cessation, but has not been studied in subjects with bipolar disorder. This 12-week open label trial will be conducted to assess the feasibility, acceptability, and safety of varenicline in bipolar depressed smokers, given in addition to the subject's primary treatment for bipolar disorder. The primary study hypothesis was that the abstinence rate for bipolar depressed patients will be 50%.

DETAILED DESCRIPTION:
Varenicline, a nicotinic acetylcholine receptor partial agonist, has been shown in two placebo-controlled trials to be efficacious for smoking cessation. Given the high prevalence of nicotine dependence in bipolar disorder and the high prevalence of sub-syndromal and syndromal depressive symptoms in bipolar disorder, this 12-week adjunctive varenicline open label trial will be conducted to assess the feasibility, acceptability, and safety of varenicline in bipolar depressed smokers. All subjects will receive individual behavioral counseling.

Primary hypothesis: the abstinence rate for bipolar depressed patients will be 50%. Secondary hypothesis: At final visit, bipolar depressed patients who have achieved remission, defined as a Montgomery Asberg Depression Rating Scale (MADRS) <8, will have a higher rate of tobacco abstinence than depressed patients who did not achieve remission (MADRS >/= 8).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 -65 years
* Meet DSM-IV criteria for bipolar disorder type I or II and nicotine dependence
* DSM-IV confirmed current major depressive episode OR current depressive symptoms defined as MADRS > 4 & <20
* Smoke at least 10 cigarettes per day
* Fagerström Test of Nicotine Dependence (FTND) score of 5 or higher
* Agree to identify collateral individuals for contact purposes to facilitate follow-up appointments
* Currently on mood stabilization treatment. A minimum daily therapeutic dosage of at least one mood stabilizer, and on the same dose for at least 2 weeks:

  * Lithium (0.6-1.2 mEq/L or 900 mg), Valproate (50-125 mg/mL or 1000 mg), Carbamazepine (4-12 mg/mL or 800 mg), Oxcarbazepine 1200 mg, Lamotrigine 100 mg, Olanzapine 10mg, Risperidone 2mg, Quetiapine 300mg, Ziprasidone 40mg, Aripiprazole 7.5 mg
  * Antidepressants are not exclusionary.
  * Topiramate is an acceptable mood stabilization treatment. There is an evidence base (Delbello et al. 2005) highlighting efficacy of topiramate monotherapy for acute mania in children and adolescents with bipolar disorder type 1.

[Mood stabilizers are a standard American Psychiatric Association (APA) treatment guidelines for Bipolar I disorder (history of mania). While the guidelines for Bipolar II disorder are unclear (history of hypomania), we feel mood stabilization provides standardization of treatment and maximizes safety (ie: preventing switch from depression to mania or hypomania).]

Exclusion Criteria:

* DSM-IV dependence for a substance other than nicotine or caffeine within past 3 months.
* DSM-IV criteria of schizophrenia or other non-affective psychotic disorder
* Psychotic symptoms within the past month
* Active suicidality as measured by screening questions from the Columbia-Suicide Severity Rating Scale (C-SSRS
* History of medically serious suicide attempt as reviewed by doctor.
* Current use (past 30 days) of other smoking cessation treatments
* Pregnant or nursing women, or women who refuse to use adequate birth control
* Serious, active or unstable medical condition
* Individuals, in the investigators opinion, unable to comply with study procedures
* Inability to provide written informed consent in English
* Allergic reaction to varenicline
* Individuals who are on dialysis or have a history of kidney disease (varenicline is excreted 96% unchanged through the kidneys) or Creatine supplementation or current anticipated daily NSAID use
* Presence of a personality disorder, that upon review of the medical record, appears to be the primary reason for psychiatric care.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Frye, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11 patients were enrolled from the community all with bipolar depression and the desire to stop smoking.
Pre-assignment Details: 36 patients who were screened did not meet inclusion/exclusion criteria and excluded from participation.
Groups:
- Varenicline: Open-label; subjects will receive a behavioral intervention in addition to Varenicline. Varenicline (Chantix®, Pfizer) is an oral medication with a recommended dosage of 0.5 mg once daily for 3 days, increasing to 0.5 mg twice daily for days 4-7, and then to the maintenance dose of 1 mg twice daily for the 12 weeks of treatment.
Period: Overall Study
Arm/Group | Varenicline
Started | 11
Completed | 5
Not Completed | 6
Not completed — Screen Failure after Consent | 2
Not completed — Adverse Event | 1
Not completed — Worsening of depression | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Varenicline
Number analyzed (Participants) | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 38.8 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 11
Brief Questionnaire of Smoking Urges (QSU-brief) [Mean (Standard Deviation); unit: Units on a scale] — The USU-brief is used as a measure of craving or desire to smoke. It uses 10 "agree-disagree" statements in a rating scale, five covering need to smoke for relief and five covering positive desire to smoke for reward. Maximum score = 1000, indicates a high level of craving. Minimum score = 0, indicates no craving for smoking. Cox LS, Tiffany ST, Christen AG. Evaluation of the brief questionnaire of smoking urges (QSU-brief) in laboaratory and clinical setting. Nicotine & Tobacco Research (2001)3(1):7-16.
  Units on a scale | 476 (89.3)
Cigarettes (per day) [Mean (Standard Deviation); unit: Cigarettes] | 15.8 (2)
Carbon Monoxide Breath Level [Mean (Standard Deviation); unit: ppm] — Measured by expired breath in parts per million (ppm). (0-10 = non smoker; 11-20 = light smoker; >20 = heavy smoker)
  ppm | 20 (4.6)
Montgomery-Asberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: Units on a scale] — MADRS is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Each item on the MADRS is scaled 0 through 6. Lowest score = 0, would indicate no depressive symptoms. Highest score = 60, indicating extreme depression. MADRS score > 20 is syndromal depression. Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry 1979; 134:382-389.
  Units on a scale | 9.9 (1.5)
Young Mania Rating Scale (YMRS) [Mean (Standard Deviation); unit: Units on a scale] — YMRS is an eleven-item, multiple choice diagnostic questionnaire which psychiatrists use to measure the severity of manic episodes in patients already diagnosed with mania. Lowest score = 0, normal subject; Highest score = 60, highly manic subject. For this scale the following scores are associated with these grades of severity: mania (YMRS = 20), hypomania (YMRS = 12), under 5 is classified as non-manic. Young RC, Biggs JT, Ziegler Ve, Meyer DA. A rating scale for mania: reliability, validity and sensitivity. BR J Psychiatry 1978; 133:429-435.
  Units on a scale | 1.9 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Carbon Monoxide Breath Level at 12 Weeks
Description: Measured by expired breath in parts per million (ppm)
Time Frame: 12 weeks
Population: Intention to Treat (ITT)
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Varenicline
Number analyzed (Participants) | 5
ppm | 6 (2.1)

2. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) at 12 Weeks
Description: MADRS is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Each item on the MADRS is scaled 0 through 6. Lowest score = 0, would indicate no depressive symptoms. Highest score = 60, indicating extreme depression. MADRS score > 20 is syndromal depression. Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry 1979; 134:382-389.
Time Frame: 12 weeks
Population: Intention to Treat (ITT)
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Varenicline
Number analyzed (Participants) | 5
Units on a Scale | 6 (2.4)

3. Secondary Outcome: Young Mania Rating Scale (YMRS) at 12 Weeks
Description: YMRS is an eleven-item, multiple choice diagnostic questionnaire which psychiatrists use to measure the severity of manic episodes in patients already diagnosed with mania. Lowest score = 0, normal subject; Highest score = 60, highly manic subject. For this scale the following scores are associated with these grades of severity: mania (YMRS = 20), hypomania (YMRS = 12), under 5 is classified as non-manic. Young RC, Biggs JT, Ziegler Ve, Meyer DA. A rating scale for mania: reliability, validity and sensitivity. BR J Psychiatry 1978; 133:429-435.
Time Frame: 12 weeks
Population: Intention to Treat (ITT)
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Varenicline
Number analyzed (Participants) | 5
Units on a Scale | 4 (1.5)

ADVERSE EVENTS:
Time Frame: 12 weeks per participant
Arm/Group | Varenicline
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 5/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=9)
Elevated blood pressure (Cardiac disorders) | 1 (1)
Compartmental Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Worsening Depression (Psychiatric disorders) | 2 (2)
Lack of concentration (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size; limitations finding participants with stable state within their bipolar disorder.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No